CLINICAL TRIAL: NCT05971875
Title: A Multinational Randomized Controlled Trial Including Two Identical Sub Studies Comparing Vaginal Versus vNOTES (Vaginal Natural Orifice Transluminal Surgery) Hysterectomy or Laparoscopic Versus vNOTES Hysterectomy.
Brief Title: RCT on 3 Types of Hysterectomy
Acronym: VANOLAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Jan Baekelandt, MD (Other)
Responsible Party: Sponsor-Investigator, Dr Jan Baekelandt, MD, Prof, Imelda Hospital, Bonheiden
Organization: Imelda Hospital, Bonheiden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vanolah
Record Dates: First submitted 2023-07-07; First posted 2023-08-02 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Minimally Invasive Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vNOTES vs Vaginal Hysterectomy (Active Comparator): Group A: If VH is concidered safe and feasable; the patient is randomized between VH and vNOTES
  Interventions: Procedure: vNOTES vs Vaginal Hysterectomy
- vNOTES vs Laparoscopic Hysterectomy (Active Comparator): If VH is not concidered safe and feasable; The patient is randomized between LH and vNOTES
  Interventions: Procedure: vNOTES vs Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: vNOTES vs Vaginal Hysterectomy — Comparison of vNOTES vs VH
  Arms: vNOTES vs Vaginal Hysterectomy
Procedure: vNOTES vs Laparoscopic Hysterectomy — Comparison of vNOTES vs LH
  Arms: vNOTES vs Laparoscopic Hysterectomy

SUMMARY:
A randomized controlled trial comparing the vaginal, vNOTES ( vaginal natural orifice transluminal surgery) or laparoscopic approach for hysterectomy in women with benign gynaecological disease

DETAILED DESCRIPTION:
Multi-center pragmatic non-blinded RCT including 1000 women 18-75 years in need of hysterectomy for benign disease; comparing VH vs vNOTES or LH vs vNOTES.

ELIGIBILITY:
Inclusion Criteria:

• Women aged 18 to 75 years regardless of parity with benign indication for hysterectomy

Exclusion Criteria:

* Women with a stage II+ prolapse in need of a hysterectomy as part of vaginal prolapse repair
* hysterectomy due to suspected endometriosis
* subtotal hysterectomy
* history of rectal surgery
* suspected malignancy
* suspected obliteration of the pouch of Douglas following severe PID or other causes
* active lower genital tract infection
* pregnancy
* failure to provide written informed consent prior to surgery
* requirement of in-patient care due to other co-morbidities

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
proportion of women leaving the hospital within 12 hours after surgery complications. | 12 hours
  Day sugery

SECONDARY OUTCOMES:
Hospitalization time | 6 weeks
  Time admitted
conversion rates | 12 hours
  conversion to different surgival technique
duration of the surgical procedure | 12 hours
  from placement of Foley to last stich
Intraoperative complications. | 12 hours
  Complication
postoperative complications, | 6 weeks
  Clavien Dindo
re-admission requiring hospitalization | 6 weeks
  Readminssion
Patient Reported Outcome Measures. | 3 months postop
  Short Female Sexual Function Index.

CONTACTS AND LOCATIONS:
Overall Officials: JAn Baekelandt, Principal Investigator — Imeldaziekenhuis
Locations (2):
- Dept of Obstetrics and Gynecology, Zadar, Croatia
- Dept of Obstetrics and Gynecology, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baekelandt JF, Stuart A, Wagenius J, Laenen A, Mol BW, Deprest J, Bosteels JJA. VaNoLaH trial: a study protocol-a multinational randomised controlled trial including two identical substudies comparing vaginal versus vNOTES (vaginal natural orifice transluminal surgery) hysterectomy or laparoscopic versus vNOTES hysterectomy. BMJ Open. 2024 Apr 23;14(4):e081979. doi: 10.1136/bmjopen-2023-081979. PMID 38658010